CLINICAL TRIAL: NCT06703294
Title: A Prospective, Multicenter, Blind, Randomized Controlled, Optimal Clinical Trial to Evaluate the Safety and Efficacy of Medical Collagen Fillers for Facial Dermal Tissue Filling to Correct Frontal Wrinkles (crow's Feet)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fiman (Changchun) Pharmaceutical Biotechnology Company Limited (Other)
Collaborators: The Seventh Medical Center of the Chinese People's Liberation Army General Hospita (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FimanPharma
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Intentional Correction of Forehead Wrinkles (crow's Feet)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Varying degrees of crow's feet (Other): Bovine collagen filling crow's feet
  Interventions: Procedure: Crow's feet injection filling; Procedure: Humanized collagen filling crow's feet

INTERVENTIONS:
Procedure: Crow's feet injection filling — Patients with crow's feet of different degree were randomly divided into two groups, which were injected with bovine collagen and humanized collagen respectively
Procedure: Humanized collagen filling crow's feet — Bovine collagen filling crow's feet

SUMMARY:
With the development of medical technology and the improvement of life treatment, people's concept of aging is also changing, people of all ages are constantly pursuing a young and healthy life, the use of lasers and fillers to correct facial wrinkles has become more and more common. For the use of fillers to correct facial wrinkles, the efficacy and safety have been fully established, to the extent that it is a minimally invasive treatment, due to its short operation time and rapid recovery, it is considered a very effective treatment for facial wrinkles.

Collagen is a kind of natural protein. As the main component of skin tissue, it has the advantages of good biocompatibility, degradability and low immunogenicity, and is an ideal material for correcting facial soft tissue defects. Collagen is implanted under the skin in a non-surgical way to increase the capacity of the dermis tissue, thus achieving the purpose of smoothing wrinkles, improving facial defects, and sculpting perfect skin. The medical collagen filling agent of Filaman (Changchun) Pharmaceutical Biotechnology Co., Ltd. consists of 3.5% bovine collagen It is composed of 0.3% lidocaine hydrochloride saline suspension, and is filled by injection to repair the shape and correct the contour to achieve satisfactory results. The product is eventually completely degraded in the human body, and the expected absorption time is 6-12 months.

In accordance with the requirements of the Medical Device Registration and Filing Management Measures, the Medical Device Clinical Trial Quality Management Standards, the Clinical Trial Registration Review Guidelines for Facial Injection Fillers (Draft for Comment), the Clinical Trial Design Guidelines for Medical devices, and the ethical principles of the Declaration of Helsinki of the World Medical Congress, To maximize the benefit of the subject and avoid as much harm as possible.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old (including 18 and 65 years old), regardless of gender; Intentional correction of forehead wrinkles (crow's feet);

Exclusion Criteria:

* Received bovine collagen fillers or hyaluronic acid within 12 months prior to enrollment

Facial area of calcium hydroxyapatite (CaHA), poly-L-lactic acid (PLLA) or plastic therapy

Domain therapy, or subjects who plan to receive such therapy during study participation;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blind investigators graded the severity of wrinkles at 1 month, 6 months, and 12 months after the last treatment Table (WSRS) score | Blind investigators graded the severity of wrinkles at 1 month, 6 months, and 12 months after the last treatment Table (WSRS) score

IPD SHARING:
Plan to Share IPD: No